CLINICAL TRIAL: NCT04347707
Title: Building Regulation in Dual Generations: Pilot Study
Brief Title: Building Regulation in Dual Generations
Acronym: BRIDGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was ended after one year due to the suspension of in-person research as a result of the COVID-19 pandemic. We have returned to the program development stage as we explore telehealth alternative options.
Sponsor: University of Manitoba (Other)
Collaborators: Research Manitoba (Other); Centre for Addiction and Mental Health (Other); University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2019:063
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Depression; Self-regulation; Child Development
Keywords: maternal mental health; self-regulatory mechanisms
MeSH Terms: conditions — Depression; Self-Control

STUDY DESIGN:
Intervention Model Description: The study will recruit a group of mother-child dyads in which the mother meets the current criteria for depression. Those mothers will participate in a 20-week group therapy intervention that incorporates Dialectical Behavior Therapy (DBT) and parent skills training. A control group of mother-child dyads who will be income and child age-matched to the intervention sample will also be recruited. These mothers will not meet the criteria for depression and will not receive the group therapy intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIDGE Clinical Group (Experimental): This group of mother-child dyads will have mothers who have been screened for and met diagnostic criteria for depression. Mothers in this group will participate in the 20-week group therapy and parent skills training intervention.
  Interventions: Behavioral: BRIDGE Therapy Program
- Baseline Comparison Group (No Intervention): This group of mother-child dyads will not meet diagnostic criteria for depression and will serve as a comparison group for baseline measures. Dyads will be matched to the BRIDGE clinical group based on household income and child age.

INTERVENTIONS:
Behavioral: BRIDGE Therapy Program — The BRIDGE Therapy Program is a novel structured form of therapy that incorporates key parenting concepts and related Dialectical Behavior Therapy (DBT) modules. The primary aim of the program is to promote self-regulation in the mother-child dyads. The program involves 20, once per week, scheduled group therapy sessions that last for 2 hours. There are two components of the program, the first is the DBT section, which will follow the DBT Skills Training Manual 2nd Edition and will target maternal mental health symptomology. The second section is the parent skill training materials, which have been designed to correspond to the 4 core DBT modules (Mindfulness, Emotion Regulation, Distress Tolerance, and Interpersonal Effectiveness) and to promote self-regulatory skill development and a positive parent-child relationship.
  Arms: BRIDGE Clinical Group

SUMMARY:
Families who experience maternal mental illness and a variety of chronic stressors are currently underserved by the parenting programs. The investigators propose that impairments in maternal self-regulation, which result in unsupportive parenting, directly impact children's own self-regulation and neurobiology, leading to risk for intergenerational transmission of mental illness. The objective of this study is to develop and evaluate a program that is targeted at improving underlying self-regulatory mechanisms in both mothers with depression and their 3 to 5-year-old children. It is hypothesized that children exposed to maternal mental illness will have greater self-regulatory deficits across emotional and behavioural domains, compared to children not exposed to mental illness. The effects of maternal mental illness are expected to be compounded for children of mothers reporting a higher degree of chronic stressors, including poverty, housing instability, violence, and low social support. Further, it is hypothesized that taking a dual-generation intervention approach to addressing self-regulatory mechanisms underlying psychopathology at the level of the mother, child, and dyad (i.e. parenting interactions) will improve both maternal capacities and child outcomes. The objectives for this study are to 1) establish a better understanding of the self-regulatory processes that are altered in preschool-aged children exposed to maternal mental illness, and determine the mediating role of parenting behaviours, as well as the moderating impact of chronic stress exposure; and 2) develop and evaluate a novel dual-generation intervention for mothers with mental illness and their 3 to 5-year-old children based on existing gold-standard evidence-based approaches.

DETAILED DESCRIPTION:
Exposure to maternal mental illness early in life can have a negative effect on children's own mental health and behavior problems putting them at risk for intergenerational transmission of mental illness (Comaskey et al., 2017; Reupert, Maybery, Nicholson, Gopfert, & Seeman, 2015; Goodman et al., 2011; O'Connor, Monk, & Burke, 2016; Dean et al., 2018; Roos et al., 2016). In order to address this concern, there have been recent calls for action for the development of early intervention programs (Shonkoff, 2016; Chartier, 2016; Patel et al., 2016; Waddell et al., 2007) that support both mother and child in a dual generation capacity (Luthar & Eisenberg, 2017; Shonkoff & Fisher, 2013). In this study, the investigators are particularly interested in the mechanisms involved in maternal self-regulation, defined as the effortful regulation of one's emotions and behaviors and what effect it has on children's self-regulation. The investigators propose that dysfunction in maternal self-regulation serves as a risk factor for the intergenerational transmission of mental illness. Partially due to the fact that dysregulation in mother's own emotions puts them at risk for mental illness and can also lead to challenges in developmentally supportive parenting (Aldao, Gee, De Los Reyes, & Seager, 2016; Kochanska, Philibert, & Barry, 2009; Strauman, 2017; Zeytinoglu, Calkins, Swingler, & Leerkes, 2017) such as scaffolding emotional socialization, stress management, impulse control (Zeytinoglu et al., 2017, Crandall, Deater-Deckard, & Riley, 2015) and often at times leads to implementation of poor parenting practices (Choi et al., 2018; Dittrich et al., 2018). Children ages 3-5 are of particular interest as they are in a developmentally sensitive period of self-regulation skills (Blair & Diamond, 2008; Gilliom, Shaw, Beck, Schonberg, & Lukon, 2002; Woodward, Lu, Morris, & Healey, 2017). The aim of this study is to gain further insight into what factors of maternal mental illness are most relevant to the development of children's self-regulatory impairments and negative outcomes. The study will also investigate how exposure to chronic stress interacts with maternal mental illness to affect development. The investigators are especially interested in studying the effects of chronic stress exposure on biological stress-related systems such as the hypothalamic-pituitary-adrenal axis (HPA) and the autonomic nervous system (ANS) to see how intervention can target these systems.

The study has two primary objectives:

1. Establish a better understanding of the self-regulatory processes that are altered in preschool-aged children exposed to maternal mental illness, and determine the mediating role of parenting behaviours, as well as the moderating impact of chronic stress exposure The investigators predict that children with mothers who have a mental illness will have more self-regulatory deficits and that this relationship will be partially mediated by parenting skills. Whereas the effects of maternal mental illness will be exacerbated by exposure to chronic stress.
2. Develop and evaluate a novel dual-generation intervention for mothers with mental illness and their 3 to 5-year-old children based on existing gold-standard evidence-based approaches. The investigators predict that our dual generation approach to intervention will improve self-regulatory outcomes in both mother and child.

Methodology

Intervention Group:

Mothers experiencing symptoms of mental illness will be recruited from the local agencies serving this population and the general community. All interested participants will be phone screened to determine eligibility. If a participant passes the phone screener questionnaire, they will be scheduled for the intake interview in which a PhD level clinical psychology graduate student will complete the MINI Neuropsychiatric Interview (Sheehan et al., 1997) to determine if the participant has experienced a recent major depressive episode. If this is found to be the case, the participant is scheduled for a 2.5 hour laboratory assessment (T1) in which mother and child will participate a variety of self-report, behavioral, and biological assessments (see primary outcome measures for more details).

After the T1 assessment, mothers will participate in the novel BRIDGE Therapy Program, which occurs once a week for 2 hours for 20 weeks. The BRIDGE Therapy Program is a mix of Dialectical Behaviour Therapy (DBT) and parent skills training. DBT aims to support clients in achieving "a life worth living" by reducing self-destructive behaviours and scaffolding self-regulatory skills while acknowledging the inherently difficult experiences individuals have endured (Valentine, Bankoff, Poulin, Reidler, & Pantalone, 2015). DBT has proven to be effective in treating a wide range of mental illnesses characterized by self-regulatory deficits (Valentine et al., 2015; Tomlinson & Hoaken, 2017; Behavioral Research & Therapy Clinics, 2018). DBT content also shares many characteristics with evidence-based interventions aimed at promoting childhood self-regulation (Maag, 2016; Bierman & Motamedi, 2015), and because of this, the parenting component of the BRIDGE Therapy program is matched to the four DBT modules; mindfulness, interpersonal effectiveness, emotion regulation, and distress tolerance. Throughout the program, data will be collected weekly on attendance, DBT/parenting skill implementation through the use of diary cards, and at weeks 2, 9, 15 on child behavior and symptoms of depression (see secondary outcome measures).

After the completion of the 20-week BRIDGE Therapy Program participants will come in for a second laboratory assessment (T2) which will follow identical procedures to those outlined in T1.

Participants will be compensated for their time at each assessment on an ascending pay scale. They will be provided with $30.00 compensation for their intake interview, $60.00 for assessment 1, and $90.00 for assessment 2. The ascending pay scale is provided to encourage retention and has been used in previous projects by the primary researcher and collaborators. Furthermore, systematic efforts will be taken to reduce barriers to treatment and encourage retainment. Participants will be aided in transportation costs (i.e. bus tickets) and provided with meals and childcare services while in group therapy sessions and for lab visits.

Control Group:

A sample of household income and age-matched mother-child dyads not exposed to maternal mental illness will be recruited and participate in identical intake and assessment (T1) procedures to the ones described above. The primary goal of the income-matched control families is to provide comparison information about baseline differences in child characteristics associated with maternal mental illness that informs the directionality of expected intervention effects.

Planned Analyses:

The investigators will examine the extent to which our measures are related using correlational analyses. The investigators will use Mplus software to examine multivariate analyses. Mother age, child age, and child gender will be examined as covariates. Child gender will also be examined as a moderator in domains that have a theoretical and evidence base.

Objective 1. When group differences emerge, structural equation models will characterize the extent to which maternal self-regulation predicts child characteristics and parenting mediates effects. Chronic stress exposure will also be examined as a moderator of associations. Objective 2.To measure the effects of the intervention repeated measure analyses will be used to examine the changes in our primary measures for mothers and children in the BRIDGE Therapy program. Next, exploratory analyses will be used to determine the extent to which changes in maternal function predict changes in each child outcome. Structural equation models will be employed to identify the relative contributions of maternal characteristics to changes in child outcomes as well as moderating (i.e. chronic stress, child gender) and mediating (i.e. parenting) paths of interest.

Expected Outcomes:

The BRIDGE Therapy Program is a novel intervention that is designed to target self-regulatory deficits and prevent the inter-generational transmission of mental illness due to these deficits. The program addresses the gaps in the literature by targeting parenting skills and both mother and child mental health outcomes. Although this is just the pilot study of the program, data from this project will be used to influence further development of the program so that outcome measures can be further improved. By taking a rapid-cycle approach to the development of materials along with the precise evaluation of the mechanisms involved, the investigators are setting the stage for the program to be adapted to meet the needs of at-risk families and to be tested in a large-scale RCT. Furthermore, by evaluating the processes involved in self-regulation for children exposed to maternal mental illness and how they respond to the intervention will inform us of how maternal mental illness impacts development. The ultimate goal of the project is to develop a dual-generation program that can prevent the intergenerational transmission of mental illness and improve outcomes for at-risk families.

ELIGIBILITY:
Inclusion Criteria:

* Must have a 3-5 year old child
* The child must not have a diagnosed developmental delay
* Must have full or joint custody of the child
* Must meet current criteria for a Major Depressive Episode
* Must be 18 years of age

Exclusion Criteria:

* Child is outside of the 3-5 year old age range
* The child has a diagnosed developmental delay
* Mother does not have full or joint custody of the child
* Mother did not meet current criteria for a Major Depressive Episode (control group)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only mothers are eligible to participate.
Enrollment: 28 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Maternal Depression from pre-intervention to post-intervention - Beck Depression Inventory | The Beck Depression Inventory will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time once again after the program is complete (approx. 20 weeks after Time 1).
  21-item self-report inventory to measure symptoms and characteristics of depression. Participants respond to statements on a 0-3 likert scale. Higher scores indicate higher depression symptoms. The highest possible score is 60 and lowest possible score is 0.
Change in Maternal Emotion Regulation pre-intervention to post-intervention - Difficulties in Emotion Regulation Scale | The Difficulties in Emotion Regulation Scale will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  18-item self-report questionnaire with 6 sub-categories to measure emotion regulation. Participants respond to items on a 5-point likert scale. Higher scores suggest more severe problems with emotion regulation. The highest possible score is 90 and the lowest possible score is 18.
Change in Parenting Stress from pre-intervention to post-intervention - Parenting Stress Index (Short form) | The Parenting Stress Index (short form) will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  36-item self-report measure filled out by parents to measure stress level within the context of parenting. Participants respond to items on a 5-point likert scale. There are 3 sub categories. Responses to each item in a sub-category are totalled and then the 3 subcategory scores are summed to represent a total stress score. Higher scores indicated higher levels of parenting stress. Normal scores fall within the 15th to 85th percentile, and scores above the 85th percentile represent clinically elevated levels of stress.

SECONDARY OUTCOMES:
Change in the Child Behaviour Checklist from pre-intervention to post-intervention | The Child Behaviour Checklist will be completed by participants at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  103-item questionnaire that asks parents to describe their child's behavioural and emotional problems within the past 2 months.
Change in Parental Sensitivity from pre-intervention to post-intervention | Parent-child interactions will be observed and video coded at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  Parent-child interactions will be video recorded after the child has participated in an acute stressor task. The interaction will be coded to measure levels of parental sensitivity using a novel coding scale.

OTHER OUTCOMES:
Change in Parent Inhibitory Control from pre-intervention to post-intervention - Exploratory Outcome | Parent inhibitory control through the stop signal task will be measured at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  Parent inhibitory control will be measured with the stop signal computer task and the effect it has on parasympathetic and sympathetic nervous activity. Participants will have 11 electrodes placed on their body to allow for recording of cardiovascular activity. They will then participate in the stop signal computer task, in which they are required to press keys on the computer keyboard in response to shapes on the screen. Participants are required to try and withhold from pressing the keys when they hear a beep. Their ability to resist their response is an indication of inhibitory control.
Change in Child Cognitive Function from pre-intervention to post-intervention - Exploratory Outcome | Child cognitive function will be assessed at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  Child cognitive function will be assessed with behavioural regulation tasks. Specifically, children will participate in the child version of the Stroop task, in which they will be required to say the opposite in response to pictures of Day/Night images and Happy/Sad faces. Additionally, they will also participate in the Head-Toes-Knees-Shoulders task, where they will be required to point to the opposite body part as instructed.
Change in Child Stress System Reactivity and Recovery from pre-intervention to post-intervention - Exploratory Outcome | Child stress system reactivity and recovery will be measured at Time 1 prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 20 weeks after Time 1).
  Child stress system reactivity will be measured through parasympathetic and sympathetic nervous system activity and salivary cortisol. Children will participate in an acute stressor task during which they will be wearing 11 electrodes on their bodies that will be recording cardiovascular activity. Salivary cortisol will also be collected immediately before the acute stressor, immediately after, and then 15, 30, and 45 minutes after.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Kaminski, MA, Study Director — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Comaskey B, Roos NP, Brownell M, Enns MW, Chateau D, Ruth CA, Ekuma O. Maternal depression and anxiety disorders (MDAD) and child development: A Manitoba population-based study. PLoS One. 2017 May 24;12(5):e0177065. doi: 10.1371/journal.pone.0177065. eCollection 2017. PMID 28542256
- [Background] Reupert, A., Maybery, D., Nicholson, J., Göpfert, M., & Seeman, M. V. (Eds.). (2015). Parental psychiatric disorder: Distressed parents and their families. Cambridge University Press.
- [Background] Goodman SH, Rouse MH, Connell AM, Broth MR, Hall CM, Heyward D. Maternal depression and child psychopathology: a meta-analytic review. Clin Child Fam Psychol Rev. 2011 Mar;14(1):1-27. doi: 10.1007/s10567-010-0080-1. PMID 21052833
- [Background] O'Connor TG, Monk C, Burke AS. Maternal Affective Illness in the Perinatal Period and Child Development: Findings on Developmental Timing, Mechanisms, and Intervention. Curr Psychiatry Rep. 2016 Mar;18(3):24. doi: 10.1007/s11920-016-0660-y. PMID 26830882
- [Background] Dean K, Green MJ, Laurens KR, Kariuki M, Tzoumakis S, Sprague T, Lenroot R, Carr VJ. The impact of parental mental illness across the full diagnostic spectrum on externalising and internalising vulnerabilities in young offspring. Psychol Med. 2018 Oct;48(13):2257-2263. doi: 10.1017/S0033291717003786. Epub 2018 Jan 14. PMID 29331151
- [Background] Roos LE, Fisher PA, Shaw DS, Kim HK, Neiderhiser JM, Reiss D, Natsuaki MN, Leve LD. Inherited and environmental influences on a childhood co-occurring symptom phenotype: Evidence from an adoption study. Dev Psychopathol. 2016 Feb;28(1):111-25. doi: 10.1017/S0954579415000322. Epub 2015 Apr 8. PMID 25851306
- [Background] Shonkoff JP. Capitalizing on Advances in Science to Reduce the Health Consequences of Early Childhood Adversity. JAMA Pediatr. 2016 Oct 1;170(10):1003-1007. doi: 10.1001/jamapediatrics.2016.1559. PMID 27548291
- [Background] Chartier, M. (2016). The Mental Health of Manitoba's Children. Manitoba Centre for Health Policy, Rady Faculty of Health Sciences, Max Rady Colledge of Medicine, University of Manitoba.
- [Background] Patel V, Chisholm D, Parikh R, Charlson FJ, Degenhardt L, Dua T, Ferrari AJ, Hyman S, Laxminarayan R, Levin C, Lund C, Medina Mora ME, Petersen I, Scott J, Shidhaye R, Vijayakumar L, Thornicroft G, Whiteford H; DCP MNS Author Group. Addressing the burden of mental, neurological, and substance use disorders: key messages from Disease Control Priorities, 3rd edition. Lancet. 2016 Apr 16;387(10028):1672-85. doi: 10.1016/S0140-6736(15)00390-6. Epub 2015 Oct 8. PMID 26454360
- [Background] Waddell C, McEwan K, Peters RD, Hua JM, Garland O. Preventing mental disorders in children: a public health priority. Can J Public Health. 2007 May-Jun;98(3):174-8. doi: 10.1007/BF03403707. PMID 17626379
- [Background] Luthar SS, Eisenberg N. Resilient Adaptation Among At-Risk Children: Harnessing Science Toward Maximizing Salutary Environments. Child Dev. 2017 Mar;88(2):337-349. doi: 10.1111/cdev.12737. Epub 2017 Feb 1. PMID 28144962
- [Background] Shonkoff JP, Fisher PA. Rethinking evidence-based practice and two-generation programs to create the future of early childhood policy. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1635-53. doi: 10.1017/S0954579413000813. PMID 24342860
- [Background] Aldao A, Gee DG, De Los Reyes A, Seager I. Emotion regulation as a transdiagnostic factor in the development of internalizing and externalizing psychopathology: Current and future directions. Dev Psychopathol. 2016 Nov;28(4pt1):927-946. doi: 10.1017/S0954579416000638. PMID 27739387
- [Background] Kochanska G, Philibert RA, Barry RA. Interplay of genes and early mother-child relationship in the development of self-regulation from toddler to preschool age. J Child Psychol Psychiatry. 2009 Nov;50(11):1331-8. doi: 10.1111/j.1469-7610.2008.02050.x. Epub 2009 Jan 12. PMID 19207629
- [Background] Strauman TJ. Self-Regulation and Psychopathology: Toward an Integrative Translational Research Paradigm. Annu Rev Clin Psychol. 2017 May 8;13:497-523. doi: 10.1146/annurev-clinpsy-032816-045012. Epub 2017 Mar 24. PMID 28375727
- [Background] Zeytinoglu S, Calkins SD, Swingler MM, Leerkes EM. Pathways from maternal effortful control to child self-regulation: The role of maternal emotional support. J Fam Psychol. 2017 Mar;31(2):170-180. doi: 10.1037/fam0000271. Epub 2016 Dec 8. PMID 27929315
- [Background] Crandall A, Deater-Deckard K, Riley AW. Maternal emotion and cognitive control capacities and parenting: A conceptual framework. Dev Rev. 2015 Jun 1;36:105-126. doi: 10.1016/j.dr.2015.01.004. PMID 26028796
- [Background] Choi KW, Houts R, Arseneault L, Pariante C, Sikkema KJ, Moffitt TE. Maternal depression in the intergenerational transmission of childhood maltreatment and its sequelae: Testing postpartum effects in a longitudinal birth cohort. Dev Psychopathol. 2019 Feb;31(1):143-156. doi: 10.1017/S0954579418000032. Epub 2018 Mar 22. PMID 29562945
- [Background] Dittrich K, Boedeker K, Kluczniok D, Jaite C, Hindi Attar C, Fuehrer D, Herpertz SC, Brunner R, Winter SM, Heinz A, Roepke S, Heim C, Bermpohl F. Child abuse potential in mothers with early life maltreatment, borderline personality disorder and depression. Br J Psychiatry. 2018 Jul;213(1):412-418. doi: 10.1192/bjp.2018.74. Epub 2018 May 24. PMID 29792587
- [Background] Blair C, Diamond A. Biological processes in prevention and intervention: the promotion of self-regulation as a means of preventing school failure. Dev Psychopathol. 2008 Summer;20(3):899-911. doi: 10.1017/S0954579408000436. PMID 18606037
- [Background] Gilliom M, Shaw DS, Beck JE, Schonberg MA, Lukon JL. Anger regulation in disadvantaged preschool boys: strategies, antecedents, and the development of self-control. Dev Psychol. 2002 Mar;38(2):222-35. doi: 10.1037//0012-1649.38.2.222. PMID 11881758
- [Background] Woodward LJ, Lu Z, Morris AR, Healey DM. Preschool self regulation predicts later mental health and educational achievement in very preterm and typically developing children. Clin Neuropsychol. 2017 Feb;31(2):404-422. doi: 10.1080/13854046.2016.1251614. Epub 2016 Nov 1. PMID 27801620
- [Background] Sheehan, D. V., Lecrubier, Y., Sheehan, K. H., Janavs, J., Weiller, E., Keskiner, A., ... & Dunbar, G. C. (1997). The validity of the Mini International Neuropsychiatric Interview (MINI) according to the SCID-P and its reliability. European Psychiatry, 12(5), 232-241.
- [Background] Valentine SE, Bankoff SM, Poulin RM, Reidler EB, Pantalone DW. The use of dialectical behavior therapy skills training as stand-alone treatment: a systematic review of the treatment outcome literature. J Clin Psychol. 2015 Jan;71(1):1-20. doi: 10.1002/jclp.22114. Epub 2014 Jul 14. PMID 25042066
- [Background] Tomlinson, M. F., & Hoaken, P. N. (2017). The Potential for a Skills-Based Dialectical Behavior Therapy Program to Reduce Aggression, Anger, and Hostility in a Canadian Forensic Psychiatric Sample: A Pilot Study. International Journal of Forensic Mental Health, 16(3), 215-226.
- [Background] Behavioral Research & Therapy Clinics. (2018). Publications. Retrieved from: http://depts.washington.edu/uwbrtc/research/publications/
- [Background] Maag, J. W. (2016). Behavior management: From theoretical implications to practical applications. Cengage Learning.
- [Background] Bierman, K. L., & Motamedi, M. (2015). Social and emotional learning programs for preschool children. Handbook of social and emotional learning: Research and practice, 135-151.
- [Background] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096
- [Background] Abidin, R. R., & Abidin, R. R. (1990). Parenting Stress Index (PSI) (p. 100). Charlottesville, VA: Pediatric Psychology Press.
- [Background] Fabes, R.A., Eisenberg, N., & Bernzweig, J. (1990).The Coping with Children's Negative Emotions Scale: Procedures and scoring. Available from authors. Arizona State University
- [Background] Achenbach, T. M. (1999). The Child Behavior Checklist and related instruments. In M. E. Maruish (Ed.), The use of psychological testing for treatment planning and outcomes assessment (pp. 429-466). Mahwah, NJ, US: Lawrence Erlbaum Associates Publishers.
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement, 1(3), 385-401.
- [Background] Chamberlain, P., & Reid, J. B. (1987). Parent observation and report of child symptoms. Behavioral Assessment.